CLINICAL TRIAL: NCT01610960
Title: Comparison of Helmet NEXT, Helmet Standard and Facemask for Noninvasive Ventilation: a Physiological Study in Healthy Volunteers
Brief Title: Comparison of Three Noninvasive Ventilation Modes: a Physiological Study in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 8937
Record Dates: First submitted 2012-05-24; First posted 2012-06-04 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Respiratory Failure; Non Invasive Ventilation on Healthy Volunteer
Keywords: Non invasive ventilation; Helmet; NEXT Helmet; Work of breathing; Intensive care
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HELMET (Active Comparator): The HELMET and HELMET NEXT modes will be tested by each patient.
  Interventions: Device: Non invasive ventilation HELMET
- Facemask (Sham Comparator): The facemask will be used by each patient.
  Interventions: Device: Non invasive ventilation facemask (Respironics)

INTERVENTIONS:
Device: Non invasive ventilation HELMET — The HELMET and HELMET NEXT modes will be tested by each patient.
  Arms: HELMET
Device: Non invasive ventilation facemask (Respironics) — The facemask Respironics (Herrsching, Germany) will be used by each patient.
  Arms: Facemask

SUMMARY:
Noninvasive ventilation (NIV) is a well established, safe, and effective technique in improving gas exchange while reducing dyspnea and inspiratory effort in patients with either hypoxemic and hypercapnic acute respiratory failure (ARF) and averts the risk secondary to endotracheal intubation.Crucial factors for NIV success, in any forms of respiratory failure, are the tolerance to the interface used and the ability of the interface to unload inspiratory-muscle. Helmet is better tolerated over time, allowing continuous application of NIV for longer periods, while face mask has been proved to be more efficient at iso-support in unloading the respiratory muscles and improving patient-ventilator synchrony. Helmet NEXT (CaStar, NIV model, Starmed, Mirandola, Italy) is a novel type of helmet with a better compliant wall, that avoid the use of armpit braces potentially improving, compared to the standard helmet, both pressurization and patient-ventilator interaction and tolerance. The objective of this study is to compare the effects of NIV delivered via face mask, standard helmet, and NEXT helmet in terms of work of breathing, patient-ventilator interaction, and comfort.

DETAILED DESCRIPTION:
16 Healthy volunteers will be enrolled. They will be ventilated with non invasive ventilation. The Work of breathing, ventilator/patient asynchrony, and ventilatory comfort produced between face mask, Helmet and NEXT helmet will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* contraindications for nasogastric tube placement
* Respiratory disease
* Pregnancy
* No French health insurance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Work of breathing | during the single visit study (day 1)
  To estimate the work of breathing, we will determine the swings in transdiaphragmatic pressure (Pdi) and the transdiaphragmatic pressure-time product (PTPdi)

SECONDARY OUTCOMES:
Ventilatory comfort | during the single visit study (day 1)
  The comfort will be assessed by a self-assessment of the patient on a visual analog scale between 0 (excellent) and 10 (discomfort).
Patient-ventilator asynchronies | during the single visit study (day 1)
  The patient-ventilator asynchronies will be assessed by the asynchronie index (number of asynchronies / number of respiratory cycles). The number of asynchronies will be assessed by the investigator, on the records of the pression curves and the respiratory outputs.
Ventilatory parameters | during the single visit study (day 1)
  The respiratory frequency and current volume will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology & Critical Care, St Eloi University Hospital, Montpellier, France

REFERENCES:
- [Derived] Vaschetto R, De Jong A, Conseil M, Galia F, Mahul M, Coisel Y, Prades A, Navalesi P, Jaber S. Comparative evaluation of three interfaces for non-invasive ventilation: a randomized cross-over design physiologic study on healthy volunteers. Crit Care. 2014 Jan 3;18(1):R2. doi: 10.1186/cc13175. PMID 24387642